CLINICAL TRIAL: NCT06037785
Title: Biobehavioral Intervention to Reduce PTSD After ICD Shock
Brief Title: Self-Management Interventions After an ICD Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: East Carolina University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Cynthia M. Dougherty, Professor, School of Nursing, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00007840; 1R21NR020967-01 (NIH)
Record Dates: First submitted 2023-09-01; First posted 2023-09-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Implantable Defibrillator User; Stress Reaction; Ptsd; Stress Management; Social Cognitive Theory
Keywords: implantable cardioverter defibrillator; ptsd; stress management
MeSH Terms: conditions — Fractures, Stress; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPSM intervention (Experimental): Heart rate self monitoring Online shock management modules
  Interventions: Behavioral: Self-Paced Self-Management (SPSM)
- usual care (No Intervention): standard observation and post-ICD shock care at each clinic that includes ICD interrogations monitored in-person or via home monitor

INTERVENTIONS:
Behavioral: Self-Paced Self-Management (SPSM) — (SPSM) consists of two components: 1) HR Self-monitoring, and 2) online Shock Management modules (N=4) with weekly telephone coaching, completed over 1 month.
  Arms: SPSM intervention

SUMMARY:
This study, "Biobehavioral Intervention to Reduce PTSD Symptoms After an ICD Shock," addresses a critical need in cardiology care by describing the feasibility and acceptability of a timely, highly promising, electronically-delivered intervention for patients who have recently received an ICD delivered shock. The study intervention and outcomes are designed to reduce anxiety, enhance return to activities of daily living (ADLs), and prevent the development of severe distress and post-traumatic stress disorder (PTSD), and ultimately promote quality of life. The study is a two-arm, embedded mixed methods, randomized trial (N=60, 30/group). The purpose is to determine feasibility and potential effects of a self-management intervention (SPSM) plus usual care (UC) compared to UC alone, delivered during the critical 1 month period after an ICD shock when distress is high. The intervention will be delivered over 1 month following an ICD shock; a 6-month follow-up will be used to assess the sustainability of intervention effects and determine if the incidence of PTSD is reduced. SPSM includes: 1) training in heart rate (HR) self-monitoring; and 2) individualized learning through 4 self-paced, web-based modules. The study interventions are delivered at a crucial time, closely after an ICD shock when stress is high, but PTSD has not yet developed. The specific aims are to: 1) examine the effects of the SPSM intervention plus UC vs. UC alone on the primary outcome of ICD shock anxiety at 1 and 6 months post-shock event, 2) describe the impact of SPSM plus UC compared to UC alone on the secondary outcomes of total daily physical activity, depression, PTSD symptoms, QOL, salivary cortisol levels, and self-efficacy and outcome expectations at 1 and 6 months post-shock event, and 3) assess feasibility, acceptability, and safety of the SPSM intervention, SDOH will be used to describe differential responses to the SPSM intervention. This study fills a significant gap in the care of patients with an ICD, through the systematic testing of a brief, novel and cost-effective intervention that provides the knowledge and skills to improve quality of life. Study findings will be used to design future larger RCTs to test intervention effectiveness for more diverse samples and settings.

ELIGIBILITY:
Inclusion Criteria:

1. ICD implant for primary or secondary prevention of sudden cardiac arrest (SCA),
2. receipt of at least 1 ICD shock, appropriate or inappropriate, one week prior to enrollment;
3. able to read, speak and write English;
4. access to online resources and telephone for study duration.

Exclusion Criteria:

1. current diagnosis of PTSD, schizophrenia or bipolar disorder;
2. Short BLESSED score >6 indicating cognitive dysfunction [73];
3. age <18 years;
4. AUDIT-C score ≥4 for alcohol use;
5. regular non-medical use of illicit drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
ICD Shock anxiety | Baseline, 1, 6 months
  Florida Shock Anxiety Scale: range 1-50, higher is higher anxiety.

SECONDARY OUTCOMES:
Total daily physical activity(steps/day) | Baseline, 1, 6 months
  Step Watch Activity Monitor, 0-unlimited number of steps. Higher is more steps.
Depression | Baseline, 1, 6 months
  PHQ-9, 0-27. Higher is higher depression.
PTSD Symptoms | Baseline, 1, 6 months
  Post-traumatic Stress Disorder Checklist PCL-5, 0-80. Higher is higher PTSD symtpoms
Quality of Life-Physical and Mental | Baseline, 1, 6 months
  PROMIS Global v 2.0, 0-50. Higher is higher qol.
Self-Efficacy Expectations | Baseline, 1, 6 months
  Self-Efficacy Expectations-SE scale, 0-60, Higher is more self-efficacy
Outcome expectation, 0-90. Higher is higher OE. | Baseline, 1, 6 months
  OE Scale
Salivary cortisol | Baseline, 1, 6 months
  Cortisol in saliva, the range in humans varies. measured in pg/ml.
Acceptability | 6 months
  Acceptability of interventions and materials measured in terms of patient burden (time to complete questionnaires & data collection, ease in understanding, implementing the intervention). These are qualitative open ended answers to questions and do not produce a number.

OTHER OUTCOMES:
Feasibility of implementing the intervention (composite outcome) | 6 months
  Feasibility will be measured using patient recruitment and contact rates (reach within 1-3 days of shock, number screened, eligible & enrolled, proportion eligible vs agree to participate). Each of these variables creates a number for the total study. They elements are added together to get a score.
Safety (composite outcome) of the intervention | 2 years of the trial
  Safety: major adverse cardiac events, including mortality (all cause and cardiac). This is measured as yes or no. Each outcome is score and the total number is summarized.
Acceptability of the intervention (composite outcome) | 6 months
  Acceptability of interventions and materials measured in terms of patient burden (time to complete questionnaires & data collection, ease in understanding, implementing the intervention). These are qualitative open ended answers to questions and do not produce a number.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Dougherty, ARNP, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
To support efforts by other researchers in replicating this study, and clinicians and healthcare systems to implement the interventions, we will 1) share the detailed study protocol, patient provider intervention materials, measures, and tools; 2) share a de-identified dataset.
Supporting Information: Study Protocol
Time Frame: 1 year after trial completion, available for up to 5 years after trial completion
Access Criteria: Contact PI
URL: https://nursing.uw.edu/profile/?pid=4318816